CLINICAL TRIAL: NCT04131452
Title: Do Women's Quality of Life, Sexual Life and Psychological State Differ Between Patients Undergoing Fresh and Frozen Embryo Transfers: a Prospective Study
Brief Title: Women's Quality of Life, Sexual Life and Psychological State in Patients Undergoing Embryo Transfers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bahceci Health Group (Other)
Collaborators: Uskudar University (Other)
Responsible Party: Principal Investigator, Mehmet Resit Asoglu, Associate professor, Bahceci Health Group
Other Study IDs: Bahceci Mehmet Asoglu
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Infertility, Female; Anxiety State; Depression; Quality of Life; Sexual Function and Fertility Disorders
MeSH Terms: conditions — Infertility, Female; Anxiety Disorders; Depression | interventions — Bays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fresh embryo transfers: those undergoing fresh embryo transfer
  Interventions: Other: Filling out the forms including IDAS-II, BAI, SF-36 and FSFI
- Frozen embryo transfers: those undergoing frozen embriyo transfer
  Interventions: Other: Filling out the forms including IDAS-II, BAI, SF-36 and FSFI

INTERVENTIONS:
Other: Filling out the forms including IDAS-II, BAI, SF-36 and FSFI — Participants will fill out certain validated forms including the expanded version of the inventory of depression and anxiety symptoms (IDAS-II), Beck Anxiety inventory (BAI), Short Form Survey (SF-36) and Female Sexual Function Index (FSFI).

SUMMARY:
Women's quality of life, sexual life and psychological state would affect the success of embryo transfer. The primary purpose of the study is to compare women's quality of life, sexual life and psychological state using validated forms between those undergoing fresh embryo transfer and those undergoing frozen embryo transfer.

DETAILED DESCRIPTION:
There are two types of embryo transfers; fresh and frozen embryo transfers. Studies have been conducted to compare success rates between fresh and frozen embryo transfers. However, most studies have not taken into consideration women's quality of life, sexual life and psychological state in comparing fresh embryo transfer with frozen embryo transfers. These all parameters are confounding factors that may influence the success of embryo transfer. The purpose of this study is to compare women's quality of life, sexual life and psychological state using validated forms between those undergoing fresh embryo transfer and those undergoing frozen embryo transfer. The following forms will be used: expanded version of the inventory of depression and anxiety symptoms (IDAS-II), Beck Anxiety inventory (BAI), Short Form Survey (SF-36) and Female Sexual Function Index (FSFI. This study can provide evidence regarding the association between women's quality of life, sexual life and psychological state and embryo transfer success.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 - 39 years
* Body mass index between 18 -3 5 kg/m2
* Anti-mullerian hormone levele >1.1 ng/ml or antral follicle count > 8
* fresh or frozen embryo transfer using middle-quality or good-quality day 3 or 5 embryos

Exclusion Criteria:

* Age below 20 or over 39 years
* Uterine malformations
* Hypo or hyperthyroidism
* Diabetes mellitus
* Previous history of psychiatric disorders
* Use of psychiatric medications
* Systemic disorders (hypertension, chronic liver/kidney/heart problems)

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population will consist of women undergoing fresh or frozen embryo transfer after assisted reproductive treatment.
Sampling Method: Probability Sample
Enrollment: 232 (Estimated)
Dates: Start 2020-01-20 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | At around 7 weeks of gestation
  Clinical pregnancy is defined as the presence of intrauterine fetal heartbeat at around 7 weeks of gestation.

SECONDARY OUTCOMES:
Implantation rate | At around 6 weeks of gestation
  Implantation is defined as presence of intrauterine gestational sac at around 6 weeks of gestation.
Live birth rate | 24 completed weeks of gestation
  Live birth is defined as at least a live birth after 24 completed weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Resit Asoglu, Ass, prof, Principal Investigator — Bahceci Health Group
Locations (1):
- Bahceci Health Group, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Skvirsky V, Taubman-Ben-Ari O, Ben Shlomo S, Azuri J, Horowitz E. Contributors to Women's Perceived Stress at the Start of Assisted Reproductive Technology. J Psychol. 2019;153(1):23-36. doi: 10.1080/00223980.2018.1471037. Epub 2018 Sep 13. PMID 30211664
- [Result] Purewal S, Chapman SCE, van den Akker OBA. Depression and state anxiety scores during assisted reproductive treatment are associated with outcome: a meta-analysis. Reprod Biomed Online. 2018 Jun;36(6):646-657. doi: 10.1016/j.rbmo.2018.03.010. Epub 2018 Mar 23. PMID 29622404